CLINICAL TRIAL: NCT06516159
Title: Validation of the MBI-C Scale in French
Acronym: MBI-C
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0323
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Subjective Cognitive Complaint; Mild Cognitive Impairment; Neuropsychiatric Symptoms
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MBI-C Scale in French
  Interventions: Diagnostic Test: MBI-C Scale in French

INTERVENTIONS:
Diagnostic Test: MBI-C Scale in French — The original version has 34 items, divided into 5 areas:
  * a reduction in motivation, interests and initiative
  * the appearance of mood disorders
  * dysregulation of impulse management
  * loss of conventions and societal norms
  * the abnormal development of strongly held beliefs and sensory experiences
  The items are rated based on the occurrence of the severity of the disorders in the previous six months on a scale of 0 to 3.
  This scale is completed by a member of the healthcare team on the basis of information collected from the relative ("informant") either in person but also by telephone The score varies between 0 and 102. The higher the score, the more psychological and behavioral symptoms are present.
  The test lasts 10 minutes.

SUMMARY:
This study aims to validate the French version of the Mild Behavioral Impairment-Checklist (MBI-C) scale, hypothetically effective for measuring behavioral symptoms in patients presenting with a subjective cognitive complaint or mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
Neuropsychiatric symptoms are common in the prodromal stage of dementia and may precede cognitive impairment. Their presence in patients without cognitive impairment, but with a subjective cognitive complaint or mild cognitive impairment (MCI), is associated with an increased risk of progression to dementia. The concept of Mild Behavioral Impairment (MBI) was developed to identify populations at risk from the early stages of the disease. MBI is characterized by long-lasting psychiatric symptoms appearing late, in patients without cognitive deficits or with MCI, and can precede dementia.

The general hypothesis is that the French version of the Mild Behavioral Impairment-Checklist (MBI-C) scale has good psychometric capabilities to correctly measure behavioral symptoms in patients with subjective cognitive complaint or MCI. The main objective is to verify the reliability and internal and external validity of the MBI-C score. Secondary objectives include studying the prevalence of MBI and determining the best cutoff for the diagnosis of MBI in patients with MBI or subjective cognitive complaint.

This is an observational, national, multicenter and cross-sectional study. It will include 170 patients (5 per scale item, or 34 items), with an inclusion period of 24 months and a total research duration of 25 months. Patients must be over 50 years old, have had subjective cognitive complaint or mild cognitive impairment for at least 6 months, and have a person who visits them at least once a week.

Validation of the MBI-C scale in French could play a crucial role in the identification and early management of neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting a subjective cognitive complaint (SCP) or mild cognitive impairment (MCI) for at least 6 months.
* Patient with a relative visiting them at least once a week.
* No opposition from the patient and his loved one

Exclusion Criteria:

* Patient presenting criteria for major neurocognitive disorder according to DSM-V criteria.
* Neuropsychiatric symptoms secondary to concomitant treatments, or to a medical or psychiatric pathology.
* Concomitant major depressive episode (DSM-V).
* Presence of concomitant pathologies preventing participation in the study (taking tests).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild cognitive impairment or subjective cognitive complaints will be recruited via memory consultations and memory day hospitals within the Memory Research and Resources Centers (CMRR); centers of excellence for the assessment and diagnosis of cognitive disorders.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Consistency for Internal validity of the Mild Behavioral Impairment-Checklist score | Baseline
  consistency will be assessed using Cronbach's alpha and McDonald's Omega coefficients.
External validation of the Mild Behavioral Impairment-Checklist score | Baseline
  Comparison of differences between the scores of the five domains of the NeuroPsychiatric Inventory-Total Questionnaire (NPI-Q) and the MBI-C.

SECONDARY OUTCOMES:
Prevalence of Mild Behavioral Impairment (MBI) in memory center patients presenting mild cognitive impairment (MCI) or a subjective cognitive complaint (SCC). | Baseline
  Percentage of patients having the 4 items of the MBI diagnostic criteria of the International Society to Advance Alzheimer's Research and Treatment (ISTAART)
Determination of the best threshold for the diagnosis of Mild Behavioral Impairment (MBI) in patients with mild cognitive impairment (MCI) or subjective cognitive complaint (SCC). | Baseline
  The best diagnostic threshold for MBI-C will be determined using the receiver operating characteristic (ROC) curve using as a reference the diagnosis by 4 items of the MBI diagnostic criteria of the ISTAART

CONTACTS AND LOCATIONS:
Overall Officials: Maria SOTO, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - University Hospital Limoges, Limoges
  - University Hospital Nice, Nice
  - University Hospital Strasbourg, Strasbourg
  - University Hospital Toulouse, Toulouse
  - Univsersity Hospital Lyon, Villeurbanne

IPD SHARING:
Plan to Share IPD: No